CLINICAL TRIAL: NCT00313001
Title: Effects of NovoLog® Mix 70/30 (Biphasic Insulin Aspart 70/30) BID and QD vs. Byetta™ Exenatide) BID on Glycemic Control: A Multicenter, 24-Week, Open-Label, Parallel Group Study in Patients With Type 2 Diabetes Mellitus Not Achieving Glycemic Targets With Metformin and a Sulfonylurea
Brief Title: Effects of Biphasic Insulin Aspart 70/30 vs. Exenatide in Type 2 Diabetes Patients Not Reaching Blood Glucose Targets on Metformin and a Sulfonylurea.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1714
Record Dates: First submitted 2006-04-08; First posted 2006-04-11 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: exenatide

SUMMARY:
This trial is conducted in the United States of America (USA). The study will compare A1C reduction achieved in patients receiving biphasic insulin aspart 70/30 once or twice daily to patients receiving exenatide twice daily. Patients enrolled in the study will be insulin naive patients who have not achieved glycemic control with metformin and sulfonylurea.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1C: At least 8%
* Patients that were never treated with insulin before
* Current therapy with metformin and a sulfonylurea.

Exclusion Criteria:

* History of recurrent, severe hypoglycemia
* Hepatic insufficiency: ALT, AST or alkaline phosphatase > 2.5 times upper limits of laboratory's normal
* Renal insufficiency: serum creatinine > 1.3 mg/dL (males) or > 1.2 mg/dL (females)
* Severe gastrointestinal disease, including gastroparesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Superiority as assessed by HbA1c reduction | at 24 weeks

SECONDARY OUTCOMES:
Safety variables
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

REFERENCES:
- [Result] Bergenstal R, Lewin A, Bailey T, Chang D, Gylvin T, Roberts V; NovoLog Mix-vs.-Exenatide Study Group. Efficacy and safety of biphasic insulin aspart 70/30 versus exenatide in subjects with type 2 diabetes failing to achieve glycemic control with metformin and a sulfonylurea. Curr Med Res Opin. 2009 Jan;25(1):65-75. doi: 10.1185/03007990802597951. PMID 19210140
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com